CLINICAL TRIAL: NCT05655169
Title: Effectiveness of Piezocision or the Combination of Piezocision and Low-level Laser Therapy on Orthodontic Tooth Movement During En-masse Retraction and the Associated Dentoalveolar Changes: A Three-arm Randomized Controlled Trial
Brief Title: Which is Better Piezosurgery or Piezosurgery With Laser in Accelerating Orthodontic Tooth Movement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UDDS-Ortho-14-2022
Record Dates: First submitted 2022-11-20; First posted 2022-12-19 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Angle Class II
MeSH Terms: conditions — Malocclusion, Angle Class II | interventions — Piezosurgery; Orthodontic Appliances, Fixed

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Piezosurgery and low-level laser therapy (Experimental): Piezocision will be applied in this group of patients using a piezosurgery knife and after six weeks of initial retraction, low-level laser therapy will be applied in this group of patients using a diode laser device.
  Interventions: Procedure: Piezosurgery and GaALAs diode laser
- Piezosurgery only (Experimental): Piezocision will be applied in this group of patients using a piezosurgery knife
  Interventions: Procedure: Piezosurgery
- Traditional treatment without acceleration (Active Comparator): In this group of patients, the en masse retraction will be conventional without any acceleration intervention.
  Interventions: Other: Fixed orthodontic appliance

INTERVENTIONS:
Procedure: Piezosurgery and GaALAs diode laser — One incision will be made between the roots of the six upper anterior teeth, and two incisions will be made between the upper canines and the second premolars. The incisions will be 5 mm long and start 4 mm apical to the interdental papilla.
  After six weeks of piezosurgery, GaALAs diode laser (wavelength: 810 nm and exposure time of 10 seconds\point) 10 seconds per point will be applied.
  Arms: Piezosurgery and low-level laser therapy
Procedure: Piezosurgery — One incision will be made between the roots of the six upper anterior teeth, and two incisions will be made between the upper canines and the second premolars. The incisions will be 5 mm long and start 4 mm apical to the interdental papilla.
  Arms: Piezosurgery only
Other: Fixed orthodontic appliance — After the levelling and alignment phase is completed, the rectangular stainless steel archwires (0.019" × 0.025") will be inserted, then after two weeks, the en masse retraction will be started via closed nickel-titanium coil springs applying 250 g of force per side.
  Arms: Traditional treatment without acceleration

SUMMARY:
Sixty patients who need extraction-based treatment of the maxillary first premolars with subsequent retraction of the maxillary anterior teeth will be divided randomly into three groups: piezocision group, piezocision with low-level laser therapy group, and control group. In each group, after the levelling and alignment phase is completed, the rectangular stainless steel archwires (0.019" × 0.025") will be inserted, then after two weeks, the en masse retraction will be started via closed nickel-titanium coil springs applying 250 g of force per side. For anchorage, mini implants will be inserted between the second premolars and the first molar on each side.

DETAILED DESCRIPTION:
Regarding the Piezocision, vertical soft-tissue incisions will be made on the buccal and palatal gingiva. One incision will be made between the roots of the six upper anterior teeth, and two incisions will be made between the upper canines and the second premolars. The incisions will be 5 mm long and start 4 mm apical to the interdental papilla. Then a piezosurgery knife will be inserted to perform the cortical alveolar incisions with 3-mm in-depth and 8 mm in length. No suturing will be needed.

Regarding the piezocision with the later application of low-level laser therapy (LLLT):

After six weeks of piezosurgery, a diode laser (wavelength: 810 nm and exposure time of 10 seconds\point) 10 seconds per point will be applied on each tooth of the six maxillary anterior teeth according to this protocol: the root will be divided theoretically into two halves; gingival and cervical, and the laser will be applied in the center of each half from both buccal and palatal sides which means four application points and total energy of 16 Joules per tooth. LLLT irradiation will be performed in the sixth week after the onset of mass retraction (day 0). After that, irradiation is repeated on days 3, 7, and 14, then every two weeks, until the class I canine relationship is achieved and/or spaces lateral to incisors are closed

ELIGIBILITY:
Inclusion Criteria:

1. Adult healthy patients, Male and female, Age range: 17-28 years.
2. Class II Division 1 malocclusion :

   * Mild/moderate skeletal Class II (sagittal discrepancy angle ≤7)
   * Overjet ≤10
   * Normal or excessive facial height (Clinically and then cephalometrically assessed using these three angles: mandibular/cranial base angle, maxillary/mandibular plane angle, and facial axis angle)
   * Mild to moderate crowding ≤ 4
3. Permanent occlusion.
4. Existence of all the upper teeth (except third molars).
5. Good oral and periodontal health:

   * Probing depth < 4 mm
   * No radiographic evidence of bone loss.
   * Gingival index ≤ 1
   * Plaque index ≤ 1

Exclusion Criteria:

1. Medical problems that affect tooth movement (corticosteroid, nonsteroidal anti-inflammatory drugs (NSAIDs), …)
2. Presence of primary teeth in the maxillary arch
3. Missing permanent maxillary teeth (except third molars).
4. Poor oral hygiene or Current periodontal disease:

   * Probing depth ≥ 4 mm
   * radiographic evidence of bone loss
   * Gingival index > 1
   * Plaque index > 1
5. The patient had previous orthodontic treatment

Ages: 17 Years to 28 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 63 (Actual)
Dates: Start 2019-10-09 (Actual); Primary Completion 2021-01-12 (Actual); Study Completion 2021-12-20 (Actual)

PRIMARY OUTCOMES:
The rate of en-masse retraction of upper anterior teeth | This will be assessed at the end of the active treatment, which is expected to occur within five months
  The rate of en-masse retraction of upper anterior teeth (mm/month) in each group will be calculated. This outcome will be measured by the following steps: Drawing a projection from the upper canine apex to the middle palatal bone line. Drawing a projection from the upper central incisor edge to the middle palatal bone line. Drawing a projection from the mesial ending of the third palatal rugae to the middle palatal bone line. Measuring the distance (mm) between the canine apex and third palatal rugae projections. Measuring the distance (mm) between the central incisor edge and third palatal rugae projections. The rate of en-masse retraction will be measured by dividing the distance between the canine apex/central incisor edge projections and the third palatal rugae projection by the time elapsed between assessment times.
Change in the anteroposterior movement of the molar | Time 0:1 day before the beginning of the retraction phase (baseline). Time 1: after 1 month from the beginning. Time 2: after 2 months. Time 3: after 3 months. Time 4: after 4 months. Time 5: immediately after the end of the retraction phase
  The anteroposterior movement of the molar (mm/month) in each group will be calculated. This outcome will be measured on the dental casts by drawing two projections from the central groove of the first maxillary molar and the mesial ending of the third palatal rugae to the middle palatal bone line. The anteroposterior movement of the first maxillary molar (mm) will be measured by dividing the distance between the two projections by the time elapsed between assessment times.
Change in the inter-canine width | Time 0:1 day before the beginning of the retraction phase (baseline). Time 1: after 1 month from the beginning. Time 2: after 2 months. Time 3: after 3 months. Time 4: after 4 months. Time 5: immediately after the end of the retraction phase
  The change in the inter-canine width (mm/month) in each group will be calculated. Assessment will be performed by measuring the distance between the cusp tips of the two upper canines. This variable will be measured on dental casts.
Change in the inter-molar width at 5 months | Time 0:1 day before the beginning of the retraction phase (baseline). Time 1: after 1 month from the beginning. Time 2: after 2 months. Time 3: after 3 months. Time 4: after 4 months. Time 5: immediately after the end of the retraction phase
  The change in the inter-molar width (mm/month) in each group will be calculated. Assessment will be performed by measuring the distance between the central groove of the two first maxillary molars. This variable will be measured on dental casts.

SECONDARY OUTCOMES:
Change in molar antero-posterior position | Time 0:1 day before the beginning of the retraction phase (baseline). Time 1: after 1 month from the beginning. Time 2: after 2 months. Time 3: after 3 months. Time 4: after 4 months. Time 5: immediately after the end of the retraction phase
  The amount of distance being travelled by the first molars is going to be measured on study models taken at monthly intervals until the end of the retraction phase.

CONTACTS AND LOCATIONS:
Overall Officials: Mudar Mohammad Mousa, DDS, Principal Investigator — Department of orthodontics, Damascus University, Syria; Mohammad Y. Hajeer, DDS,MSc,PhD, Study Director — Department of orthodontics, Damascus University, Syria
Locations (1):
- University of Damascus, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abdelhameed AN, Refai WMM. Evaluation of the Effect of Combined Low Energy Laser Application and Micro-Osteoperforations versus the Effect of Application of Each Technique Separately On the Rate of Orthodontic Tooth Movement. Open Access Maced J Med Sci. 2018 Nov 15;6(11):2180-2185. doi: 10.3889/oamjms.2018.386. eCollection 2018 Nov 25. PMID 30559886
- [Background] Alfawal AMH, Hajeer MY, Ajaj MA, Hamadah O, Brad B, Latifeh Y. Evaluation of patient-centered outcomes associated with the acceleration of canine retraction by using minimally invasive surgical procedures: A randomized clinical controlled trial. Dent Med Probl. 2020 Jul-Sep;57(3):285-293. doi: 10.17219/dmp/120181. PMID 32909702
- [Background] Hatrom AA, Zawawi KH, Al-Ali RM, Sabban HM, Zahid TM, Al-Turki GA, Hassan AH. Effect of piezocision corticotomy on en-masse retraction. Angle Orthod. 2020 Sep 1;90(5):648-654. doi: 10.2319/092719-615.1. PMID 33378476
- [Background] Al-Ibrahim HM, Hajeer MY, Alkhouri I, Zinah E. Leveling and alignment time and the periodontal status in patients with severe upper crowding treated by corticotomy-assisted self-ligating brackets in comparison with conventional or self-ligating brackets only: a 3-arm randomized controlled clinical trial. J World Fed Orthod. 2022 Feb;11(1):3-11. doi: 10.1016/j.ejwf.2021.09.002. Epub 2021 Oct 21. PMID 34688577
- [Background] Khlef HN, Hajeer MY, Ajaj MA, Heshmeh O, Youssef N, Mahaini L. The effectiveness of traditional corticotomy vs flapless corticotomy in miniscrew-supported en-masse retraction of maxillary anterior teeth in patients with Class II Division 1 malocclusion: A single-centered, randomized controlled clinical trial. Am J Orthod Dentofacial Orthop. 2020 Dec;158(6):e111-e120. doi: 10.1016/j.ajodo.2020.08.008. Epub 2020 Nov 4. PMID 33158633
- [Derived] Mousa MM, Hajeer MY, Alam MK, Aljabban O, Almahdi WH. Evaluation of low-level laser therapy and piezocision in the en-masse retraction of upper anterior teeth. Eur J Orthod. 2025 Apr 8;47(3):cjaf026. doi: 10.1093/ejo/cjaf026. PMID 40353446